CLINICAL TRIAL: NCT01930656
Title: The Effectiveness of Using Mobile Device and the World Health Organization Fracture Risk Assessment Tool (FRAX®) to Assist Osteoporosis Assessment and Management
Brief Title: Mobile Device to Help FRAX® Screening
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201208029RIC
Record Dates: First submitted 2013-07-03; First posted 2013-08-29 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Osteoporosis; Fracture
Keywords: osteoporisis; fracture; risk; cost effectiveness; FRAX; mobile device
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group A, B, C: Group A- American cut-point Group B- Translational approach cut-point Group C- Cost-effectiveness cut-point

SUMMARY:
Background: The Taiwanese FRAX® (Fracture Risk Assessment Tool) calculator is available online for clinical use. Our Taiwanese Osteoporosis Clinical Treatment Guidelines suggests using the American high risk cut-points for considering treatment but also suggests deriving domestic cut-points from cost-effective approach. Establishing cost-effective domestic cut-points for policy suggestions coupled with mobile devices with wireless access would potentially increase the usage of FRAX® tool.

Objectives: 1) Using literature review to establish cost-effectiveness FRAX® cut-points. 2) To assess the effectiveness of mobile devices assisted FRAX® tool based osteoporosis diagnostic and management model. 3) To provide FRAX® based reimbursement policy suggestions.

Methods: 1) Investigators will use FRAX®, cost-effectiveness and other key words to search Pubmed and international osteoporosis guidelines to better understand the clinical applications of FRAX® in other countries. Investigators will also search epidemiological data for osteoporosis, facture, quality of life and cost to establish domestic cost-effeteness, and translational approach FRAX® cut-points. 2) Three targeting populations from National Taiwan University Hospital (NTUH) are selected for prospective study (Group A: geriatric health exam clinics with American cut-points, group B: orthopedic clinics with translational approach cut-points and group C: endocrine clinics with cost-effectiveness cut-points,). A mobile device with app application coupled with the FRAX® tool is used by a trained research assistant during clinic waiting periods to screen and enroll high risk (75 from each clinic) adults with informed consents. Participants are referred to geriatric clinics for systemic osteoporosis diagnoses and managements. Percentage of participants that meet the current NHI medication reimbursement regulation and percentage of self-pay medications are calculated. Analysis is stratified by age and gender. 3) The impacts of 3 different cut-points on increment NHI reimbursement are estimated. An osteoporosis expert group meeting is to be held for FRAX® based osteoporosis medication reimbursement modifications to the NHI and the Department of Health.

Expected Outcomes: 1) To establish the mobile device assisted FRAX® based osteoporosis screening and management model. 2) Base on the study results and expert consensus, investigators will provide policy suggestions of FRAX® based reimbursement modifications.

DETAILED DESCRIPTION:
This is an observational study. The study outcomes might base on clinical physician opnions to provide policy suggestion of FRAX® at which cut-point is considering for treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 40-90
* screen high risk from FRAX

Exclusion Criteria:

* treated with anti-osteoporosis medications within last 3-12 months (depends on medication types)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults visitng geraitric health exam clinics, orthopedic clinic, and endocrinology clinic
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of enrollment cases | in 6 month
  target 75 in each group, total 225

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan